CLINICAL TRIAL: NCT04253093
Title: Comparison of Rocuronium Induced Neuromuscular Blockade in Late Second Trimester Pregnant and Non-pregnant Women
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hallym University Kangnam Sacred Heart Hospital (Other)
Responsible Party: Principal Investigator, Choi Eun MI, professor, Hallym University Kangnam Sacred Heart Hospital
Other Study IDs: 2019-05-008
Record Dates: First submitted 2020-01-29; First posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Pregnancy Related

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The present study is to compare the onset and duration of rocuronium in late second trimester women and non-pregnant women undergoing general anesthesia.

DETAILED DESCRIPTION:
Pregnancy induces physiological changes. Plasma volume, cardiac output, hepatic blood flow and protein binding are changed from the first trimester of pregnancy. These physiological changes give effect to the onset and duration of neuromuscular blocking drugs.

Rocuronium is a commonly used neuromuscular blocking drug categorized as FDA category B. Rocuronium is widely used for pregnant women. Previous studies have evaluated the onset and duration of rocuronium in postpartum women. Lately, the investigators have evaluated the onset and duration of rocuronium in early second trimester pregnant women and the duration was significantly longer in early second trimester women compared to non-pregnant women.

Since there is little research on the onset and duration of rocuronium in the late second trimester pregnant women, the investigators planned the present research.

ELIGIBILITY:
Inclusion Criteria:

* women undergoing general anesthesia

Exclusion Criteria:

* liver disease
* renal disease
* diabetes mellitus
* asthma
* allergic to specific drugs
* BMI>30 or <18

Ages: 20 Years to 45 Years | Sex: Female
Age Groups: Adult
Study Population: case: late second trimester pregnant women undergoing general anesthesia control: non-pregnant women undergoing general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-10-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
duration of rocuronium | time measured to 25% recovery with T1 using Train of Four watch, assessed upto 1 hour
  time measured with TOFwatch-SX

SECONDARY OUTCOMES:
onset of rocuronium | time measured to 0% depression of T1 using Train of Four watch, assessed upto 5 minutes
  time measured with TOFwatch-SX

CONTACTS AND LOCATIONS:
Overall Officials: Eunmi Choi, Study Chair — professor
Locations (1):
- Kangnam sungshim hospital, Seoul, South Korea